CLINICAL TRIAL: NCT00833144
Title: Emergency Physician-Performed Thoracic Ultrasound Rapidly Identifies Patients With Congestive Heart Failure
Brief Title: Bedside Ultrasound Identifies Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Sierra Beck, MD, RDMS, Assistant Professor, Emory University
Other Study IDs: IRB00015895; 2008125 (Other: Other)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Heart Failure; Dyspnea
Keywords: heart failure; dyspnea; ultrasound
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Congestive Heart Failure
- 2: Patients without congestive heart failure

SUMMARY:
Patients often arrive to the Emergency Department with the chief complaint of shortness of breath. The cause of the shortness of breath may be due to many things, such as pneumonia, emphysema, a heart attack, heart failure, and others. It is often very difficult for the physician to determine the cause of the shortness of breath in the first two hours in the Emergency Department. This ambiguity makes treating the patient very difficult. Although a patient could benefit from treatment upon arrival, the emergent treatment of the condition must wait until a final diagnosis is made.

Recently, emergency physicians have been using portable ultrasound at the patient's bedside to diagnose numerous conditions, including trauma, blood clots, kidney stones, etc. Recent research suggests that heart failure, one of the causes of shortness of breath, may be diagnosed within 5 minutes or less using ultrasound. Most of these studies come from the intensive care and cardiology. However, no research has yet been performed to determine if emergency physicians can effectively use ultrasound to quickly diagnose and treat heart failure within the first few minutes of a patient's arrival to the emergency department. The hypothesis of this study is to evaluate the ability of residents in emergency medicine to use ultrasound to diagnose patients in heart failure who presented with the chief complaint of shortness of breath. The final diagnosis of the patient upon discharge from the hospital will be compared to the preliminary diagnosis based on the portable ultrasound findings.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* presenting complaint of shortness of breath or dyspnea

Exclusion Criteria:

* prisoners
* pregnant women
* shortness of breath clearly secondary to another diagnosis (i.e. trauma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Care Center with the chief complaint of shortness of breath or dyspnea will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of the ultrasound lung rockets to predict congestive heart failure | One year

SECONDARY OUTCOMES:
comparison of the BNP with the thoracic ultrasound findings | One year

CONTACTS AND LOCATIONS:
Overall Officials: William Manson, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Agricola E, Bove T, Oppizzi M, Marino G, Zangrillo A, Margonato A, Picano E. "Ultrasound comet-tail images": a marker of pulmonary edema: a comparative study with wedge pressure and extravascular lung water. Chest. 2005 May;127(5):1690-5. doi: 10.1378/chest.127.5.1690. PMID 15888847
- [Background] Jambrik Z, Monti S, Coppola V, Agricola E, Mottola G, Miniati M, Picano E. Usefulness of ultrasound lung comets as a nonradiologic sign of extravascular lung water. Am J Cardiol. 2004 May 15;93(10):1265-70. doi: 10.1016/j.amjcard.2004.02.012. PMID 15135701
- [Background] Lichtenstein D, Meziere G. A lung ultrasound sign allowing bedside distinction between pulmonary edema and COPD: the comet-tail artifact. Intensive Care Med. 1998 Dec;24(12):1331-4. doi: 10.1007/s001340050771. PMID 9885889
- [Background] Maisel AS, Krishnaswamy P, Nowak RM, McCord J, Hollander JE, Duc P, Omland T, Storrow AB, Abraham WT, Wu AH, Clopton P, Steg PG, Westheim A, Knudsen CW, Perez A, Kazanegra R, Herrmann HC, McCullough PA; Breathing Not Properly Multinational Study Investigators. Rapid measurement of B-type natriuretic peptide in the emergency diagnosis of heart failure. N Engl J Med. 2002 Jul 18;347(3):161-7. doi: 10.1056/NEJMoa020233. PMID 12124404